CLINICAL TRIAL: NCT06678009
Title: The Effect of 8-week Isokinetic Training Combined with Blood Flow Restriction on Muscle Strength and Endurance in Runners
Brief Title: Isokinetic Training Combined with Blood Flow Restriction on Muscle Strength and Endurance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bihter Aslanyurek (Other)
Responsible Party: Sponsor-Investigator, Bihter Aslanyurek, Associate Professor Ph.D, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Gulhane; 321S398 (Other Grant/Funding Number: Scientific and Technological Research Council of Türkiye)
Record Dates: First submitted 2024-11-04; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Blood Flow Restriction
Keywords: blood flow restriction (BFR); isokinetic training

STUDY DESIGN:
Intervention Model Description: A total of 42 runners were randomly assigned to either the isokinetic training group with blood flow restriction (BFR Group; n= 21) or the isokinetic training group without blood flow restriction (Control Group; n= 21).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The isokinetic training group with blood flow restriction (BFR Group) (Active Comparator): For the BFR, the occlusion pressure was set to 80% of arterial occlusion pressure as determined. The isokinetic training protocol for the knee flexor and extensor muscles consisted of 3 sets of 10 repetitions in 60°/sec and 3 sets of 30 repetitions in 180°/sec for 8 weeks, 2 times per week for 16 sessions.
  Interventions: Device: the isokinetic training group with blood flow restriction
- The isokinetic training group without blood flow restriction (Control Group) (Other): The isokinetic training group without blood flow restriction. The isokinetic training protocol for the knee flexor and extensor muscles consisted of 3 sets of 10 repetitions in 60°/sec and 3 sets of 30 repetitions in 180°/sec for 8 weeks, 2 times per week for 16 sessions
  Interventions: Device: the isokinetic training group without blood flow restriction

INTERVENTIONS:
Device: the isokinetic training group with blood flow restriction — The isokinetic training protocol for the knee flexor and extensor muscles consisted of 3 sets of 10 repetitions in 60°/sec and 3 sets of 30 repetitions in 180°/sec for 8 weeks, 2 times per week for 16 sessions.
  Arms: The isokinetic training group with blood flow restriction (BFR Group)
Device: the isokinetic training group without blood flow restriction — The isokinetic training protocol for the knee flexor and extensor muscles consisted of 3 sets of 10 repetitions in 60°/sec and 3 sets of 30 repetitions in 180°/sec for 8 weeks, 2 times per week for 16 sessions.
  Arms: The isokinetic training group without blood flow restriction (Control Group)

SUMMARY:
Evidence regarding the effectiveness of blood flow restriction during isokinetic exercises is insufficient. When the literature is reviewed, it is seen that there are very few studies investigating the effect of isokinetic training program with blood flow restriction on muscle strength and endurance in healthy athletes. In line with this information, the aim of this study was to investigate the effect of an 8-week isokinetic training program combined with blood flow restriction on knee flexor and extensor maximal muscle strength and endurance in runners.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effect of lower extremity isokinetic training combined with blood flow restriction (BFR) on knee flexor and extensor muscle strength and endurance in runners. A total of 42 runners were randomly assigned to either the isokinetic training group with blood flow restriction (BFR Group; n= 21) or the isokinetic training group without blood flow restriction (Control Group; n= 21). For the BFR, the occlusion pressure was set to 80% of arterial occlusion pressure as determined. The isokinetic training protocol for the knee flexor and extensor muscles consisted of 3 sets of 10 repetitions in 60°/sec and 3 sets of 30 repetitions in 180°/sec for 8 weeks, 2 times per week for 16 sessions. The muscle strength and endurance were evaluated before and after the training program using an isokinetic dynamometer.

ELIGIBILITY:
Inclusion Criteria: the absence of heart disease, arterial hypertension, diabetes mellitus or any musculoskeletal condition of the lower extremities that precluded participation in the recommended training protocols and testing, no use of any dietary supplements during the study and for at least 2 months prior to the study and running more than 20 kilometers per week.

-

Exclusion Criteria: Age <20 or >40, history of cardiac disease, history of heart failure, history of coronary artery disease, history of peripheral artery disease, presence/history of varicose veins, history of hypertension, history of diabetes mellitus, history of pulmonary disease, history of pulmonary embolism, history of hematological disease, history of previous deep vein thrombosis, pregnancy, use of oral contraceptives, use of anticoagulants, history of previous surgery in the lower extremity, body mass index >25, history of cancer, presence of lymphedema, history of lymphadenectomy, history of trauma in the lower extremity within the last 6 months or 1 year.

-

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of lower extremity muscle strength and muscular endurance using isokinetic dynamometry in runners who met the inclusion criteria for the study. | Baseline and 8 weeks
  Isokinetic knee flexor and extensor muscles strength and endurance were evaluated with the isokinetic dynamometer. All the athletes underwent twice a week for 8 weeks of isokinetic training protocol. Both groups performed the same isokinetic training protocol. Blood flow restriction was applied to the BFR group while the athletes doing isokinetic training protocol, but not to the control group. Isokinetic knee flexor and extensor muscles strength and endurance were re- evaluated at the end of the intervention (48 hours after the last training session).

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin F. Çetinkaya, MD, Study Director — Gulhane Training and Research Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - University of Health Sciences, Gulhane Faculty of Medicine, Ankara, Ankara
  - Bihter Akınoğlu, Ankara

IPD SHARING:
Plan to Share IPD: Yes
Supporting information (data) will be shared once it is available for publication.
Supporting Information: Study Protocol, CSR
Time Frame: Supporting information will be shared once it is available for publication.
Access Criteria: Supporting information will be uploaded to the journal in which it is submitted for publication.